CLINICAL TRIAL: NCT04699773
Title: Laser Interstitial Thermal Therapy Followed By Hypofractionated Radiation Therapy For Treatment Of Newly Diagnosed High-Grade Gliomas
Brief Title: LITT Followed by Hypofractionated RT for Newly Diagnosed Gliomas (GCC 20138)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Keep Punching Foundation (Unknown)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00094285
Record Dates: First submitted 2021-01-04; First posted 2021-01-07 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Glioma; Glioblastoma; Brain Tumor
Keywords: Laser Interstitial Thermal Therapy; Brain Tumor; Radiotherapy; Proton Therapy; Glioma
MeSH Terms: conditions — Glioma; Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- LITT with Hypofractionated RT (Experimental): Laser interstitial thermal therapy (LITT) followed by hypo-fractionated radiation therapy, 25Gy/10 fractions.
  Interventions: Procedure: LITT; Radiation: Hypofractionated Radiation Therapy

INTERVENTIONS:
Procedure: LITT — This procedure is done under MRI guidance and employs low-powered thermal energy to achieve tumor ablation through coagulation.
  Other Names: Laser Interstitial thermal therapy
Radiation: Hypofractionated Radiation Therapy — Treatments will be delivered once daily on consecutive treatment days (typically 5 fractions per week). Radiation therapy simulation is to be performed within 10 days of the LITT procedure.

SUMMARY:
The purpose of this study is to evaluate the treatment regimen of using Laser Interstitial Thermal Therapy (LITT) and Hypo-fractionated Radiation Therapy to treat patients with newly diagnosed gliomas.

DETAILED DESCRIPTION:
Radiation therapy is preferably used as an adjunct to surgery for patients with a newly diagnosed or recurrent glioblastoma. LITT offers an alternative to surgical resection, and due to its minimally invasive nature, does not delay initiating radiation therapy. Another advantage of LITT prior to radiation therapy is the ability to obtain a tissue diagnosis of the tumor prior to initiating radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with radiographic evidence of suggestive of a primary high-grade glioma
2. Brain MRI with contrast demonstrates an enhancing mass within 60 days prior to registration. Patient must be deemed a candidate for LITT from MRI by Neurosurgery in order to be eligible.
3. History and physical including neurological exam within 30 days prior to registration
4. Karnofsky performance status ≥50% within 30 days prior to registration
5. Age ≥ 18 years old
6. Patients must have signed an approved informed consent
7. Patients with the potential for pregnancy or impregnating their partner must agree to practice effective contraceptive methods to avoid conception while on study and for 6 months after study completion.
8. Female patients of child-bearing potential must have a negative pregnancy test within 28 days prior to study registration.

Exclusion Criteria:

1. Patients that are not surgical candidates for stereotactic biopsy or laser ablation
2. Patients with impaired cardiac function or clinically significant cardiac diseases, including any of the following:

   * History or presence of serious uncontrolled ventricular or significant arrhythmias.
   * Any of the following within 6 months prior to registration: myocardial infarction, severe/unstable angina, coronary artery bypass graft, congestive heart failure, cerebrovascular accident, transient ischemic attack , pulmonary embolism
3. Infratentorial tumor or evidence of leptomeningeal spread
4. Inability to undergo a MRI
5. Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 2 years
  The ability to complete protocol treatment (i.e. LITT and radiation therapy) without undue treatment-related acute toxicity as defined below:
  * Safety: < 40% rate of irreversible Grade 3 or higher neurologic treatment-related toxicity
  * Early stopping rules: Two or more Grade 2 or higher symptomatic CNS hemorrhages; Eight treatment-related Grade 3 or higher non-hematologic or Grade 4 or higher hematologic treatment related toxicities

SECONDARY OUTCOMES:
Progression-free survival at 6 months | 6 months
  To describe progression-free survival rate in subjects with newly diagnosed high-grade gliomas treated with Laser Interstitial Thermal Therapy
Median progression-free survival | 2 years
  To describe median progression-free survival rate in subjects with newly diagnosed high-grade gliomas treated with Laser Interstitial Thermal Therapy followed by hypofractionated radiation therapy.
Median overall survival | 2 years
  To describe median progression-free survival rate in subjects with newly diagnosed high-grade gliomas treated with Laser Interstitial Thermal Therapy followed by hypofractionated radiation therapy.
1-year overall survival | 1 year
  To describe 1- year survival rate in subjects with newly diagnosed high-grade gliomas treated with Laser Interstitial Thermal Therapy followed by hypofractionated radiation therapy.
Overall response rate | 2 years
  To describe overall response rate in subjects with newly diagnosed high-grade gliomas treated with Laser Interstitial Thermal Therapy followed by hypofractionated radiation therapy.
Quality of Life assessed by M.D. Anderson Symptom Inventory | 2 years
  Patient reported quality of life impact from undergoing LITT followed by hypofractionated radiation therapy using the M.D. Anderson Symptom Inventory- Brain Tumor (MDASI-BT) questionnaire.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - UCH Kaufman Cancer Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology, Columbia, Maryland
  - Baltimore Washington Medical Center, Glen Burnie, Maryland

IPD SHARING:
Plan to Share IPD: No